CLINICAL TRIAL: NCT04830007
Title: Factors Associated With the Absence of Contraception at the Time of Unplaned Pregnancy Among Women Seeking a Voluntary Termination of Pregnancy
Brief Title: Factors Associated With the Absence of Contraception at Women Seeking a Voluntary Termination of Pregnancy
Status: Suspended | Type: Observational
Why Stopped: Investigator coordinatoor left the site and the trial
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: NOCONTRAIVG; 2021-A00298-33 (Other: ID-RCB)
Record Dates: First submitted 2021-02-11; First posted 2021-04-02 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy, Unwanted
Keywords: Contraception; Abortion; Unplanned pregnancy; Unintended pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be offered to all women who are consultant for an abortion plan are seen in consultation at the orthogeny center where the study will be conducted. Of these 700 women, about 10% will not agree to participate in the study and 10% will not meet the inclusion criteria. Thus it's plane to include 560 patients in the study.

DETAILED DESCRIPTION:
In 1967, the Neuwirth law allowed women to control their fertility by establishing the right to contraception as a principle. Since then, they have continued to take ownership of the various contraceptive methods, which are regularly renewed.

Contraceptive coverage is important in France as it is estimated that 92% of women of childbearing age use a contraceptive method. The pill remains the most widely used method of contraception (36.5%), ahead of the intrauterine device (25.6%) condoms (15.5%) Several laws have been introduced from 1967 to today to facilitate access to sexual health care: screening for sexually transmitted infections, free provision of emergency contraception to minors, non-prescription delivery of emergency contraception, free consultation at a family planning and education center, voluntary termination of pregnancy 100%, reimbursement of condoms by social security.

Despite all the measures put in place, it is now clear that the number of unplanted pregnancies is decreasing slightly and the number of abortion has remained stable since 2001.

According to the latest literature data, several socio-demographic factors appear to play a role in the rate of use of voluntary termination of pregnancy., including age, socio-cultural level, marital and economic status and ethnic origin. All the more striking, it appears that while voluntary termination of pregnancy are mainly related to contraceptive failures, one third of them involve women who do not have contraception. According to the latest Ined survey, and in accordance with other data from the literature, the factors associated with the absence of contraceptive use are multiple: ignorance about fertility, family or cultural context, cost of contraceptive methods or lack of information related to them.

While these studies have looked at the reasons given by women for the lack of contraception, with little data on the characteristics of these women, particularly socio-demographics and their reproductive history and in particular in the context of unwanted pregnancy. This finding leads us to question the factors associated with the absence of contraception among women in demand of a voluntary termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* woman of 18 years of age or older;
* Being French-speaking;
* request for a medical or instrumental voluntary termination of pregnancy
* No opposition to participation in the protocol
* Be affiliated with a social security plan

Exclusion Criteria:

* desired pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregant women
Study Population: Protocol proposed to woman who wanted a voluntary termination of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Association between absence of contraception and socio-demographic factors, characteristics of pregnancy abortion and medical follow-up | 1 hour
  Statistically significant association between the absence of contraception in patients consulting for a voluntary termination of pregnancy and socio-demographic factors, characteristics of voluntary termination of pregnancy abortion and characteristics related to medical follow-up

SECONDARY OUTCOMES:
Prescription and dispensing of contraception | 1 hour
  Prevalence of patients informed about the prescription and dispensing of contraception including emergency contraception
Existence of family planning centers | 1 hour
  Prevalence of patients informed about the existence of family planning centers
Emergency contraception | 1 hour
  Prevalence of women who have used emergency contraception
Price and reimbursement of condoms | 1 hour
  Prevalence of women informed about the price and reimbursement of condoms
Knowledge of conception | 1 hour
  Estimate the percentage of women who thought they could get pregnant at the time of the intercourse that led to this pregnancy
Fertile window | 1 hour
  Prevalence of women who use a method to track their fertile window
Affection of fertility | 1 hour
  Estimate the percentage of women who think that contraception can affect their fertility

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Villeneuve St Georges, Villeneuve-Saint-Georges, France